CLINICAL TRIAL: NCT04982159
Title: Correlation Between Minimum Inhibitory Concentration and Clinical Outcome of Invasive Fusariosis
Status: Completed | Type: Observational
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Other Study IDs: FIB-VOR-2019-01
Record Dates: First submitted 2021-07-06; First posted 2021-07-29 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Invasive Fusariosis
Keywords: invasive fusariosis; minimum inhibitory concentration
MeSH Terms: conditions — Fusariosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Invasive Fusariosis: Patients hospitalized with an invasive fusariosis diagnostic in the stablished period of study.
  Interventions: Other: There is no intervention. This is an observational study.

INTERVENTIONS:
Other: There is no intervention. This is an observational study. — There is no intervention. This is an observational study.

SUMMARY:
Multi-centered, international, observational and retrospective study to analyze the correlation between MIC and clinical outcome in patients with invasive fusariosis.

ELIGIBILITY:
Inclusion Criteria:

* Invasive fusariosis diagnostic
* Proof of anti-fungic susceptibility according to EUCAST or CLSI, for the medicine used in the treatment of invasive fusariosis.
* Available data about anti-fungic medicines used: name of medicine, start and end date of treatment.
* Available information about clinical outcome of illness after 30 days, 6 weeks and 90 days (dead or alive).
* Only cases of invasive fusariosis proven or possible will be included.

Exclusion Criteria:

* None

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Hospital patients diagnosed with invasive fusariosis.
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical Evolution | 6 weeks after diagnosis
  Retrospective evaluation of death rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Reina Sofía, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared after the study concludes and results are published.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: When study is published.
Access Criteria: Through request to Principal Investigator.
URL: https://pubmed.ncbi.nlm.nih.gov/33326585/